CLINICAL TRIAL: NCT02664701
Title: Cognitive Behavioural Group Therapy Versus Individual Supportive Therapy for the Prevention of Repeat Suicide Attempts: a Multicentre, Assessor-blinded, 2-parallel-group, Randomised, Superiority Trial
Brief Title: Cognitive Behavioural Group Therapy Versus Individual Supportive Therapy for the Prevention of Repeat Suicide Attempts
Acronym: G-PACTS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHRC-N/2014/MA-01; 2015-A01585-44 (Other: RCB number)
Record Dates: First submitted 2016-01-19; First posted 2016-01-27 (Estimated); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Suicidal Ideation; Suicide, Attempt
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual supportive therapy (Active Comparator): Patients randomized to this arm will have individual supportive therapy.
  Intervention: Baseline evaluation with a psychiatrist
  Intervention: Individual supportive therapy
  Intervention: Evaluations with a psychiatrist
  Interventions: Other: Baseline evaluation with a psychiatrist; Other: Individual supportive therapy; Other: Evaluations with a psychiatrist
- Cognitive behavioural group therapy (Experimental): Patients randomized to this arm will have cognitive behavioural therapy.
  Intervention: Baseline evaluation with a psychiatrist
  Intervention: Cognitive behavioural group therapy
  Intervention: Evaluations with a psychiatrist
  Interventions: Other: Baseline evaluation with a psychiatrist; Other: Cognitive behavioural group therapy; Other: Evaluations with a psychiatrist

INTERVENTIONS:
Other: Baseline evaluation with a psychiatrist — Baseline data and questionnaires are established.
Other: Individual supportive therapy — 6 sessions of individual supportive therapy with a psychologist, 1 session per week for 6 weeks
  Arms: Individual supportive therapy
Other: Cognitive behavioural group therapy — 6 sessions of cognitive behavioural group therapy with a psychologist, 1 session per week for 6 weeks
  Arms: Cognitive behavioural group therapy
Other: Evaluations with a psychiatrist — Evaluation withs a psychiatrist in the 10 days following the end of psychotherapy, then at 3, 6, 9, and 12 months.

SUMMARY:
The primary objective of this study is to evaluate the efficacy of a program of 6 sessions of Cognitive Behavioural Group Therapy (CBGT) (as compared to 6 sessions of Individual Supportive Therapy (IST)) designed for preventing repeat suicide attempts at 12 months post-psychotherapy in adults admitted to inpatient care for suicide attempts.

DETAILED DESCRIPTION:
The secondary objectives of this study are to assess the efficacy of CBGT on:

A. parameters describing the incidence of suicide and repeat suicide attempts, as well as suicide re-attempt free follow-up time,

B. long-term changes in suicidal ideation,

C. long-term changes in psychiatric symptoms (depression, hope for the future, hospitalization).

ELIGIBILITY:
Inclusion Criteria:

* The patient has been correctly informed
* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* French speaking adults (18 years or older) freely hospitalized (in centres or via emergency services) for prevention of suicide and who have a medium or high suicide risk score according to a Mini International Neuropsychiatric Interview structured interview
* Presence of suicidal ideation according to the Beck Suicide Ideation Scale (score > 3)
* Prior (or recent) suicide attempt within the last three month
* The patient is able to understand the study and capable of giving his/her informed consent
* The patient is available during the weekly time slots proposed by the investigator

Exclusion Criteria:

* The patient is participating in another study that may interfere with the results or conclusions of this study
* Within the past three months, the patient has participated in another study that may interfere with the results or conclusions of this study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, or is an adult under guardianship
* The patient refuses to sign the consent, or it is impossible to correctly inform the patient
* Emergency situations preventing proper study conduct
* History of schizophrenia or other psychotic troubles
* Presence of psychotic symptoms at initial interview
* Serious cognitive impairment
* Medical incapacity to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2017-10-17 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
The primary clinical endpoint is the duration (in days) of a suicide reattempt-free follow-up period | 12 months

SECONDARY OUTCOMES:
The Columbia suicide severity rating scale (C-SSRS) | baseline
The Columbia suicide severity rating scale (C-SSRS) | in the 10 days after the end of psychotherapy
The Columbia suicide severity rating scale (C-SSRS) | 3 months
The Columbia suicide severity rating scale (C-SSRS) | 6 months
The Columbia suicide severity rating scale (C-SSRS) | 9 months
The Columbia suicide severity rating scale (C-SSRS) | 12 months
Completed suicide (yes/no) | in the 10 days after the end of psychotherapy
Completed suicide (yes/no) | 3 months
Completed suicide (yes/no) | 6 months
Completed suicide (yes/no) | 9 months
Completed suicide (yes/no) | 12 months
Number of suicide re-attempts during the follow-up period. | in the 10 days after the end of psychotherapy
  A suicide attempt is defined as either an "actual attempt" or an "interrupted attempt" using the definitions in the C-SSRS assessment.
Number of suicide re-attempts during the follow-up period. | 3 months
  A suicide attempt is defined as either an "actual attempt" or an "interrupted attempt" using the definitions in the C-SSRS assessment.
Number of suicide re-attempts during the follow-up period. | 6 months
  A suicide attempt is defined as either an "actual attempt" or an "interrupted attempt" using the definitions in the C-SSRS assessment.
Number of suicide re-attempts during the follow-up period. | 9 months
  A suicide attempt is defined as either an "actual attempt" or an "interrupted attempt" using the definitions in the C-SSRS assessment.
Number of suicide re-attempts during the follow-up period. | 12 months
  A suicide attempt is defined as either an "actual attempt" or an "interrupted attempt" using the definitions in the C-SSRS assessment.
Beck Suicide Ideation Scale (BSSI) | Baseline
Beck Suicide Ideation Scale (BSSI) | in the 10 days after the end of psychotherapy
Beck Suicide Ideation Scale (BSSI) | 3 months
Beck Suicide Ideation Scale (BSSI) | 6 months
Beck Suicide Ideation Scale (BSSI) | 9 months
Beck Suicide Ideation Scale (BSSI) | 12 months
Beck Depression Inventory-II (BDI-II) | Baseline
Beck Depression Inventory-II (BDI-II) | in the 10 days after the end of psychotherapy
Beck Depression Inventory-II (BDI-II) | 3 months
Beck Depression Inventory-II (BDI-II) | 6 months
Beck Depression Inventory-II (BDI-II) | 9 months
Beck Depression Inventory-II (BDI-II) | 12 months
Beck Hopelessness Scale (BHS) | Baseline
Beck Hopelessness Scale (BHS) | in the 10 days after the end of psychotherapy
Beck Hopelessness Scale (BHS) | 3 months
Beck Hopelessness Scale (BHS) | 6 months
Beck Hopelessness Scale (BHS) | 9 months
Beck Hopelessness Scale (BHS) | 12 months
Cumulative days of hospitalization | in the 10 days after the end of psychotherapy
Cumulative days of hospitalization | 3 months
Cumulative days of hospitalization | 6 months
Cumulative days of hospitalization | 9 months
Cumulative days of hospitalization | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mocrane Abbar, MD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (9):
- France (9):
  - CHU de Clermont Ferrand - Hôpital Gabriel-Montpied, Clermont-Ferrand
  - CHU de Lyon - Groupement Hospitalier Edouard Herriot, Lyon
  - CHRU de Montpellier - Hôpital Lapeyronie, Montpellier
  - Clinique Les Sophoras, Nîmes
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - CMME, Paris
  - CH Henri Laborit, Poitiers
  - CHRU de Tours - Clinique Psychiatrique Universitaire, Saint-Cyr-sur-Loire
  - CHRU de Strasbourg - Hôpital Civil, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Chaib LS, Lopez-Castroman J, Abbar M. Group Post-Admission Cognitive Therapy for Suicidality vs Individual Supportive Therapy for the prevention of repeat suicide attempts: a randomized controlled trial. Trials. 2020 Oct 27;21(1):889. doi: 10.1186/s13063-020-04816-y. PMID 33109271